CLINICAL TRIAL: NCT00143559
Title: Haploidentical Hematopoietic Stem Cell Transplantation Utilizing Partial T-Cell Depletion as Immunotherapy for Hematologic Malignancies
Brief Title: Stem Cell Transplantation as Immunotherapy for Hematologic Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: G. Hale, Principal Investigator, St. Jude Children's Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HAPREF
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2009-01-29 (Estimated); Status verified 2009-01

CONDITIONS: Leukemia; Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia; Chronic Myeloid Leukemia; Juvenile Myelomonocytic Leukemia; Myelodysplastic Syndrome; Paroxysmal Nocturnal Hemoglobinuria; Hodgkin's Lymphoma; Non-Hodgkin Lymphoma
Keywords: Allogeneic stem cell transplantation; Haploidentical stem cell transplant; Mismatched family member stem cell donor transplant; Bone marrow transplant; High risk hematological malignancies; T-cell depletion methodology; Miltenyi Biotec CliniMACS stem cell selection device
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myelomonocytic, Juvenile; Myelodysplastic Syndromes; Hemoglobinuria, Paroxysmal; Hodgkin Disease; Lymphoma, Non-Hodgkin | interventions — Antibodies; Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other)
  Interventions: Drug: Systematic chemotherapy and antibodies; Procedure: Allogeneic stem cell transplantation; Device: Miltenyi CliniMACS

INTERVENTIONS:
Drug: Systematic chemotherapy and antibodies — Systemic chemotherapy and antibodies as follows:
  Transplant recipients received a reduced intensity conditioning regimen consisting of OKT-3, fludarabine, thiotepa, and melphalan followed by an infusion of a T-cell depleted haploidentical hematopoietic stem cell graft. The antibody Rituximab was administered within 24 hours of the infusion in an effort to prevent PTLPD. In addition to T -cell depletion of the donor product, Mycophenylate mofetil was provided over several months as prophylaxis for GVHD
Procedure: Allogeneic stem cell transplantation — An infusion of HLA mismatched family member donor stem cells processed through the use of the investigational Miltenyi Biotec CliniMACS device
Device: Miltenyi CliniMACS — Miltenyi Biotec CliniMACS stem cell selection device
  Other Names: Haploidentical donor stem cell transplant; Mismatched family member transplant; Allogeneic stem cell transplant; Reduced intensity conditioning regimen; Hematopoietic stem cell transplant

SUMMARY:
Blood and marrow stem cell transplant has improved the outcome for patients with high-risk hematologic malignancies. However, most patients do not have an appropriate HLA (immune type) matched sibling donor available and/or are unable to identify an acceptable unrelated HLA matched donor through the registries in a timely manner. Another option is haploidentical transplant using a partially matched family member donor.

Although haploidentical transplant has proven curative in many patients, this procedure has been hindered by significant complications, primarily regimen-related toxicity including GVHD and infection due to delayed immune reconstitution. These can, in part, be due to certain white blood cells in the graft called T cells. GVHD happens when the donor T cells recognize the body tissues of the patient (the host) are different and attack these cells. Although too many T cells increase the possibility of GVHD, too few may cause the recipient's immune system to reconstitute slowly or the graft to fail to grow, leaving the patient at high-risk for significant infection.

For these reasons, a primary focus for researchers is to engineer the graft to provide a T cell dose that will reduce the risk for GVHD, yet provide a sufficient number of cells to facilitate immune reconstitution and graft integrity. Building on prior institutional trials, this study will provide patients with a haploidentical graft engineered to specific T cell target values using the CliniMACS system. A reduced intensity, preparative regimen will be used in an effort to reduce regimen-related toxicity and mortality.

Two groups of patients were enrolled on this study. One group included those with high-risk hematologic malignancies and the second group included participants with refractory hematologic malignancies or undergoing a second transplant. The primary aim of the study was to estimate the relapse rate in the one group of research participants with refractory hematologic malignancies or those undergoing second allogeneic transplant. Both groups will be followed and analyzed separately in regards to the secondary objectives.

This study was closed to accrual on April 2006 as it met the specific safety stopping rules regarding occurrence of severe graft vs. host disease. Although this study is no longer open to accrual, the treated participants continue to be followed as directed by the protocol.

DETAILED DESCRIPTION:
Secondary outcome evaluations for this clinical study included the following:

* To estimate one-year overall survival for research participants with high risk malignancies who receive a haploidentical HSCT
* To compare overall survival and cumulative incidence of relapse for the two groups of patients with their corresponding historical controls
* To estimate disease-free survival and event-free survival in participants with hematologic malignancies who receive a haploidentical HSCT
* To estimate the incidence of overall grade 3-4 acute GvHD in research participants with hematologic malignancies who receive a haploidentical HSCT
* To estimate the incidence of chronic GvHD and graft failure in research participants with hematologic malignancies who receive a haploidentical HSCT
* To estimate the incidence of non-hematologic regimen-related toxicity and regimen-related mortality in the first 100 days post-transplant in research participants with hematologic malignancies who receive a haploidentical HSCT
* To estimate the number of research participants who develop evidence of EBV reactivation or post-transplant lymphoproliferative disease (PTLPD)
* To describe disease-free survival, GvHD and engraftment in research participants receiving grafts from Killer immunoglobulin-like receptor (KIR) mismatched and KIR matched haploidentical donors

ELIGIBILITY:
Inclusion Criteria:

Eligible participants were assigned to one of two different strata dependent on diagnosis, disease status and/or past transplant experience. Both strata received the same intervention but will be followed and analyzed separately.

* Group A must have one of the following diagnosis

  * Acute lymphoid leukemia (ALL) in second or subsequent remission or high risk in first remission
  * Acute myeloid leukemia (AML) in remission or with ≤ 25% blasts in bone marrow
  * Chronic myeloid leukemia (CML)
  * Juvenile myelomonocytic leukemia (JMML)
  * Myelodysplastic syndrome (MDS)
  * Paroxysmal nocturnal hemoglobinuria (PNH)
  * Hodgkin's (HD) or non-Hodgkin's lymphoma (NHL) in second or subsequent remission after autologous HSCT, or unable to have hematopoietic stem cells collected for autologous HSCT
* Group B must have one of the following refractory diagnosis (chemoresistant relapse or primary induction failure)

  * Acute lymphoid leukemia (ALL)
  * Acute myeloid leukemia (AML) ≥ 25% blast in bone marrow
  * Secondary AML / MDS
  * Chronic myeloid leukemia (CML) in accelerated phase or blast crisis
  * Juvenile myelomonocytic leukemia (JMML)
  * Myelodysplastic syndrome (MDS)
  * Hodgkin's (HD) or non-Hodgkin's lymphoma (NHL) with residual disease followed by autologous HSCT or who have chemo-resistant disease
  * Or patients who have undergone prior allogeneic HSCT or who have a co-morbid condition that in the medical opinion of the Transplant Faculty makes standard myeloablation prohibited
* At least 2 and less than or equal to 21 years of age
* Lacks suitable HLA-identical sibling or matched available unrelated donor and has a mismatched family member donor that is available, HIV negative and at least 18 years old
* Cardiac shortening fraction ≥ 25%
* Creatinine clearance ≥ 40 cc/min/1.73m^2
* FVC ≥ 40% of predicted or pulse oximetry ≥ 92% on room air
* Direct bilirubin ≤ 3 mg/dL or SGPT ≤ 500 U/L
* Karnofsky or Lansky (age dependent) performance score of ≥ 50

Exclusion Criteria:

* Known allergy to murine products
* Lactating (female patient)
* Pregnancy (female patient)
* Active central nervous system (CNS) leukemia

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2005-08; Primary Completion 2006-07 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
To measure the rate of disease relapse by six months posttransplant in children and young adults with refractory hematologic malignancies who receive a haploidentical stem cell graft processed using the investigational CliniMACS cell sorting device. | September 2006

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Hale, M.D., Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org